CLINICAL TRIAL: NCT04947371
Title: Adjuvant Therapy With Anlotinib Hydrochloride for Patients With Hepatocellular Carcinoma Who Underwent Curative Resection: a Single Arm Study
Brief Title: Adjuvant Therapy With Anlotinib for HCC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The standard of care of adjuvant therapy for liver cancer was changed.
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Hui-Chuan Sun, Professor of Surgery, Shanghai Zhongshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC-ANO-ADJ
Record Dates: First submitted 2021-06-09; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; anlotinib; adjuvant; surgery
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib Hydrochloride (Experimental): Oral anlotinib 12 mg/d
  Interventions: Drug: Anlotinib Hydrochloride

INTERVENTIONS:
Drug: Anlotinib Hydrochloride — Oral anlotinib hydrochloride 12 mg/d
  Other Names: AL3818

SUMMARY:
Patients with high risk of disease recurrence after curative resection for hepatocellular carcinoma (HCC) deserve active intervention. However, there's limited treatment choice for these patients. Anlotinib hydrochloride, a multitarget tyrosine kinase inhibitor for both tumor angiogenesis and proliferative signaling in cancer cells, is approved in China for the 3rd line treatment of advanced non-small cell lung cancer. In the current study, we are to evaluate the safety and effects of adjuvant anlotinib therapy for the patients who underwent curative resection for HCC with high risk of tumor recurrence, which is defined by Shanghai Score (Sun, et al. Chin Med J (Engl) 2017).

DETAILED DESCRIPTION:
Patients with high risk of disease recurrence after curative resection for hepatocellular carcinoma (HCC) deserve active intervention. However, there's limited treatment choice for these patients. Anlotinib hydrochloride, a multitarget tyrosine kinase inhibitor for both tumor angiogenesis and proliferative signaling in cancer cells, is approved in China for the 3rd line treatment of advanced non-small cell lung cancer. In the current study, we are to evaluate the safety and effects of adjuvant anlotinib therapy for the patients who underwent curative resection for HCC with high risk of tumor recurrence, which is defined by Shanghai Score (Sun, et al. Chin Med J (Engl) 2017).

The primary outcome of this study is treatment safety, and the secondary outcome is recurrence-free survival and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18-75 years.
* HCC diagnosis was confirmed by pathological examination and those who did not receive anti-tumor treatment (anti-tumor treatment including but not limited to: local ablation therapy, TACE, radiation therapy, chemotherapy, targeted drug therapy, immunotherapy, and etc.)
* Underwent curative resection for HCC with high risk of tumor recurrence, which was defined by Shanghai Score ≥ 4.922 (Sun, et al. Chin Med J (Engl) 2017)
* Child-Pugh class: A or B7
* The ECOG Performance Status: 0-1 points
* The expected survival time ≥ 6 months
* No disease recurrence 4-6 weeks after surgery as evaluated by abdominal contrast-enhanced CT/MRI and chest CT.
* Adequate organs function
* Complete blood counting HB ≥ 90 g/L ANC ≥ 1.5×10^9 /L PLT ≥ 75×10^9/L
* Blood biochemistry ALB ≥ 28 g/L ALT and AST< 5×ULN TBIL ≤ 2×ULN Serum creatinine ≤ 1×ULN
* Women of childbearing age must have pregnancy tests within 7 days prior to admission, and the results are negative and are willing to use appropriate methods of contraception at 8 weeks after the trial and at the end of the trial. For men, surgical sterilization should be applied, or consent to use appropriate methods of contraception 8 weeks after the trial and at the end of the trial.
* Subjects voluntarily participated in the study, signed informed consent, good compliance in drug therapy and followed up.

Exclusion Criteria:

* Cholangiocarcinoma, the combination of cholangiocarcinoma of HCC, or fibrolamellar HCC diagnosed by pathology examination.
* Past or current diagnosed with other malignancy, except skin basal cell carcinoma and cervical carcinoma in situ.
* Those treated with liver or other organ transplantation or willing to undergo liver transplantation.
* The conditions not suitable for oral medications, including difficulty swallowing, chronic diarrhoea, or bowel obstruction.
* Vascular events within 6 months, including stroke and transient ischemic attack

  , deep venous thrombosis or pulmonary artery embolism.
* Alimentary tract hemorrhage or high risk of alimentary tract hemorrhage due to esophageal varices, active ulcerative lesions or ulcerative colitis; or fecal occult blood test ≥ ++, or for those with fecal occult blood test (+), gastroscopy is required.
* Abnormal coagulation function (international normalized ratio > 2, prothrombin time > 16 s, thrombin time >21s, activated partial thromboplastin time > 21 s, or fibrinogen < 2 g/L); or other conditions with bleeding tendency or undergoing thrombolysis or anticoagulant therapy.
* Other severe or uncontrolled comorbidities:
* hypertension and the blood pressure was not well managed by medications (systolic pressure ≥ 150 mmHg or diastolic pressure ≥ 90 mmHg); level 2 or higher myocardial ischemia or myocardial infarction, uncontrolled arrhythmia (including QTc interval ≥ 480 ms); level 1 heart dysfunction; or LVEF < 50%.
* active or uncontrolled infection.
* uncontrolled diabetes (fasting blood glucose > 10 mmol/L).
* Urinary protein ≥ ++ or 24 hours urine protein > 1 g.
* Unhealed wounds, ulcer, or bone fracture.
* Those with mental illness or a history of psychotropic substance abuse; HIV infection.
* Other conditions that the investigators considered that not suitable for trial inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Adverse events rate | 12 months
  The rates of severity and seriousness of the adverse events. Adverse events are graded according to the NCI-CTCAE (Version 5.0)

SECONDARY OUTCOMES:
Recurrence-free survival | 24 months
  From the date of liver surgery to the date of diagnosis of tumor recurrence or death from any cause
Overall survival | 24 months
  From the date of liver surgery to the date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Jia Fan, MD&PhD, Principal Investigator — Fudan University; Hui-Chuan Sun, MD&PhD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Han B, Li K, Wang Q, Zhang L, Shi J, Wang Z, Cheng Y, He J, Shi Y, Zhao Y, Yu H, Zhao Y, Chen W, Luo Y, Wu L, Wang X, Pirker R, Nan K, Jin F, Dong J, Li B, Sun Y. Effect of Anlotinib as a Third-Line or Further Treatment on Overall Survival of Patients With Advanced Non-Small Cell Lung Cancer: The ALTER 0303 Phase 3 Randomized Clinical Trial. JAMA Oncol. 2018 Nov 1;4(11):1569-1575. doi: 10.1001/jamaoncol.2018.3039. PMID 30098152
- [Background] Sun HC, Xie L, Yang XR, Li W, Yu J, Zhu XD, Xia Y, Zhang T, Xu Y, Hu B, Du LP, Zeng LY, Ouyang J, Zhang W, Song TQ, Li Q, Shi YH, Zhou J, Qiu SJ, Liu Q, Li YX, Tang ZY, Shyr Y, Shen F, Fan J. Shanghai Score: A Prognostic and Adjuvant Treatment-evaluating System Constructed for Chinese Patients with Hepatocellular Carcinoma after Curative Resection. Chin Med J (Engl). 2017 Nov 20;130(22):2650-2660. doi: 10.4103/0366-6999.218019. PMID 29133751